CLINICAL TRIAL: NCT00858728
Title: Effect of Fruit and Vegetable Consumption on Immune Function in the Elderly: a Randomised Controlled Trial
Brief Title: Effect of Fruit and Vegetable Consumption on Immune Function in the Elderly
Acronym: ADIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06/NIR03/64
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Immune Function
Keywords: Natural killer cell cytotoxicity; Antibody response; Tetanus toxoid vaccination; Pneumovax II vaccination; Total serum immunoglobulins; IgG subclasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5 portions fruit and vegetables/day
  Interventions: Behavioral: 5 portions
- 2 (Other): 2 portions fruit and vegetables/day
  Interventions: Behavioral: 2 portions

INTERVENTIONS:
Behavioral: 5 portions — Subjects randomised to the intervention group will be provided with a selection of fruit and vegetables once a week (from a local supermarket) and will be asked to consume 5 portions of fruit and vegetables per day. For the purposes of this study, a portion will be as defined by the Food Standards Agency, i.e. an 80 g serving (one apple, orange or banana, or 3 heaped tablespoons of vegetables).
  Arms: 1
Behavioral: 2 portions — Subjects randomised to the control group will be provided with a selection of fruit and vegetables once a week (from a local supermarket) and will be asked to consume 2 portions of fruit and vegetables per day. For the purposes of this study, a portion will be as defined by the Food Standards Agency, i.e. an 80 g serving (one apple, orange or banana, or 3 heaped tablespoons of vegetables).
  Arms: 2

SUMMARY:
The immune system undergoes a range of changes as individuals become elderly. These may manifest as an increasing susceptibility to infection or a tendency to develop autoimmune or malignant disease. Multiple underlying factors contribute to this phenomenon of immunological aging, and in this study the investigators will examine the possibility that inadequate diet may be one such contributing factor. Fruit and vegetable intake, which can be low in the elderly, is associated with reduced chronic disease risk. This proposal will test the hypothesis that increased fruit and vegetable intake may positively affect clinically relevant measures of immune function. One hundred healthy volunteers aged 65-85 years following a low fruit and vegetable diet (<=2 portions/d) will be recruited and randomised to continue following their normal diet, or to consume at least 5 portions of fruit and vegetables daily for 16 weeks. Immune function and biochemical markers of nutritional status will be assessed before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85 years
* Habitual consumption of fruit and vegetables <= 2 portions daily

Exclusion Criteria:

* Those on special diets, taking nutritional supplements or medications known to affect immune function or absorption of nutrients
* Excessive alcohol consumption (>28 U/week men or >21 U/week women)
* BMI>35 kg/m2
* History of diabetes or dementia
* Pneumovax II vaccination within previous 2 years
* Inability to provide informed consent
* Any other problem which would prevent adherence to a high fruit and vegetable diet
* Recent infection (<3 weeks since completion of any antibiotic course or symptoms of viral illness)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in natural killer cell cytotoxicity and antibody response to Tetanus toxoid and Pneumovax II vaccination | 16 weeks

SECONDARY OUTCOMES:
Change in other markers of immune function | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jayne V Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Co Antrim, United Kingdom

REFERENCES:
- [Derived] Neville CE, McKinley MC, Draffin CR, Gallagher NE, Appleton KM, Young IS, Edgar JD, Woodside JV. Participating in a fruit and vegetable intervention trial improves longer term fruit and vegetable consumption and barriers to fruit and vegetable consumption: a follow-up of the ADIT study. Int J Behav Nutr Phys Act. 2015 Dec 18;12:158. doi: 10.1186/s12966-015-0311-4. PMID 26684653
- [Derived] Neville CE, Young IS, Gilchrist SE, McKinley MC, Gibson A, Edgar JD, Woodside JV. Effect of increased fruit and vegetable consumption on physical function and muscle strength in older adults. Age (Dordr). 2013 Dec;35(6):2409-22. doi: 10.1007/s11357-013-9530-2. Epub 2013 Apr 2. PMID 23543264
- [Derived] Gibson A, Edgar JD, Neville CE, Gilchrist SE, McKinley MC, Patterson CC, Young IS, Woodside JV. Effect of fruit and vegetable consumption on immune function in older people: a randomized controlled trial. Am J Clin Nutr. 2012 Dec;96(6):1429-36. doi: 10.3945/ajcn.112.039057. Epub 2012 Nov 7. PMID 23134881